CLINICAL TRIAL: NCT02087072
Title: COLLABORATIVE HOME VISITS TO REDUCE HOSPITAL READMISSIONS AND IMPROVE MEDICATION USE DURING TRANSITIONS OF CARE
Status: Withdrawn | Type: Observational
Sponsor: Ohio State University (Other)
Collaborators: American Society of Health-System Pharmacy Foundation (Unknown)
Responsible Party: Principal Investigator, Stuart Beatty, Assistant Professor of Clinical Pharmacy, Ohio State University
Other Study IDs: 2013H0185
Record Dates: First submitted 2014-03-12; First posted 2014-03-14 (Estimated); Last update posted 2022-09-30 (Actual); Status verified 2022-09

CONDITIONS: Transitional Care Coordination; Home Visits
Keywords: home visits; transitions of care; pharmacist
MeSH Terms: interventions — Pharmacists

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Recently discharged homebound patients
  Interventions: Other: Collaborative visit with provider and pharmacist

INTERVENTIONS:
Other: Collaborative visit with provider and pharmacist

SUMMARY:
The primary objective is to develop a sustainable practice model emphasizing home visits by a collaborative physician and pharmacist team to decrease unplanned emergency department visits and hospital readmissions at 30 and 90 days for high-risk home bound patients. Secondary objectives include (1) tracking the number, type, and severity of adverse drug events (ADE) and potential adverse drug events (pADE) that occur following hospital discharge and (2) resolving any identified ADE and pADE within 7 days of hospital discharge.

Adult patients will be scheduled for a home visit by the Healthy at Home Columbus program at the time of hospital discharge. The home visit will occur within 7 days of hospital discharge and will consist of a complete hospital and medication review by a physician or nurse practitioner and a pharmacist (including all lab tests, imaging studies, medication changes, and proposed plan of care at the time of discharge). The investigators hypothesize these home visits will reduce 30 and 90 days hospital readmission rates and ED visits.

The number of emergency department visits and unplanned hospital readmissions will be tracked at 30 and 90 days following discharge from the hospitalization that led to study enrollment. A comparison cohort of patients discharged in the 12 months prior to study initiation will be used to compare the effectiveness of the home visit program. The number and type of adverse drug events (ADE) and potential adverse drug events (pADE) that occur during transitions of care will also be characterized. All ADE and pADE will be resolved during the initial home visit and will be classified based on severity. All ADE and pADE will be evaluated independently by two pharmacist reviewers; each reviewer will independently assign a severity rating to each ADE and pADE.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients discharged from the hospital in the last 7 days and with more than two chronic conditions and significant obstacles to accessing care in an office setting are eligible for study participation

Exclusion Criteria:

* Adult patients able to access care in an office setting.
* Adult patients discharged from the hospital greater than 7 days prior to the office visit.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will be selected from the OSU Healthy at Home program that have been recently discharged from the hospital.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2013-10; Primary Completion 2014-12 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
Hospital Readmission | 30 days

SECONDARY OUTCOMES:
Emergency Department Visit | 30 days

OTHER OUTCOMES:
Number of drug related problems identified | 30 days
Type of drug related problems identified | 30 days

CONTACTS AND LOCATIONS:
Locations (1):
- The Ohio State University Division of General Internal Medicine Martha Morehouse, Columbus, Ohio, United States